CLINICAL TRIAL: NCT02054117
Title: Association Between Haptoglobin Genotype and the Development of Perihematomal Edema After Spontaneous Intracerebral Hemorrhage
Brief Title: Association Between Haptoglobin Genotype and Brain Swelling
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator is leaving institution.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 201300797
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: Hemorrhage; Intracerebral hemorrhage (ICH)
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intracerebral Hemorrhage: Spontaneous intracranial or intraparenchymal hemorrhage that occurred in a supratentorial location.
  Interventions: Other: Intracerebral Hemorrhage

INTERVENTIONS:
Other: Intracerebral Hemorrhage — Spontaneous intracranial or intraparenchymal hemorrhage that occurred in a supratentorial location.
  Other Names: Spontaneious intracranial hemorrhage; Intraparenchymal hemorrhage

SUMMARY:
Intracerebral hemorrhage is bleeding into the brain and is a major cause of stroke and other complications. Brain injury from intracerebral hemorrhage occurs in two phases. The early phase involves the mechanical compression of brain tissue by the expanding hematoma. In a later phase, brain swelling develops causing further compression that may lead to brain herniation and death. This study investigates the neuroprotective role of haptoglobin, in minimizing the development of brain swelling following intracerebral hemorrhage.

DETAILED DESCRIPTION:
Intracerebral hemorrhage is bleeding into the brain parenchyma. It is a major cause of stroke, and is associated with significant morbidity and mortality. Brain injury from intracerebral hemorrhage occurs in two phases. The early phase involves the mechanical compression of brain tissue by the expanding hematoma. In a later phase, brain edema, especially perihematomal edema, develops causing further compression that may lead to brain herniation and death. Several factors are implicated in the development of brain edema, including inflammation resulting from the oxidative stress caused by iron-rich hemoglobin released from lysed erythrocytes in brain tissue. This study investigates the neuroprotective role of an acute phase reactant, haptoglobin, in minimizing the development of perihematomal edema following intracerebral hemorrhage. This protein protects brain tissue from hemoglobin degradation products by forming haptoglobin-hemoglobin complexes that are subsequently cleared by the spleen. Notably, different alleles of haptoglobin exist in humans, with varying affinities for hemoglobin. Investigating the association between the different alleles and the degree of perihematomal edema formation is the primary goal of this study. The investigators will also look at a marker of inflammation, matrix metalloproteinases, and analyze its level of expression in subjects with different alleles of haptoglobin.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracranial or intraparenchymal hemorrhage
* 18-85 years of age
* Hemorrhage occurred in a supratentorial location

Exclusion Criteria:

* Inability to obtain consent within 3 days of hemorrhage onset
* Known pregnancy
* Therapeutic anticoagulation with Lovenox, Coumadin or Heparin
* Prior history of therapeutic radiation to any area
* Brain tumor
* Hemorrhage related to trauma, aneurysm, arteriovenous malformation or other vascular malformation
* Central nervous system infection
* Subdural hematoma
* Subarachnoid hemorrhage
* Chronic immunosuppression, including steroids or chemotherapy agents
* Infratentorial location
* Unable to obtain MRI due to mental status or other contraindication (metal, pacemaker, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from within the hospital setting.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Perihematomal Edema Volume | Post-hemmorhage day 3
  Perihematomal edema will be measured by averaging the edema area over multiple slices and subtracting the hemorrhage area from the total lesion area.

CONTACTS AND LOCATIONS:
Overall Officials: Spiros Blackburn, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States